CLINICAL TRIAL: NCT01300663
Title: Creating and Validating a Patient-reported Outcome Instrument to Assess Symptom Experience Related to Surgical Wounds in Women With Vulvar Neoplasms - A Mixed Methods Study
Brief Title: A New Patient Reported Outcome Instrument to Assess Symptom Experience in Women With Vulvar Neoplasms (WOMAN-PRO)
Acronym: WOMAN-PRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Foundation Cancer Research Switzerland (Unknown)
Responsible Party: Prof. Dr. Rebecca Spirig, Institute of Nursing Science, University of Basel
Other Study IDs: 412-09; KFS 02456-08-200 (Other Grant/Funding Number: Foundation Cancer Research Switzerland, KFS 02456-08-200)
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Women With Vulvar Intraephitelial Neoplasia or Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- post-surgery symptom experience: women with vulvar intraephitelial neoplasia or vulvar cancer

SUMMARY:
Post-surgery complications in women with vulvar neoplasms (vulvar intraepithelial neoplasia and vulvar cancer) are still high and an instrument assessing patients self-reported post-vulval surgery symptom experiences is missing. The study aims to develop and validate a postoperative instrument to assess symptom experiences in women with vulvar neoplasms. In this mixed-method project 20 patients were interviewed, a WOMAN-PRO instrument was developed and content validity was tested by 6 experts and 10 patients. The instrument's psychometric properties and the prevalence of symptoms will be examined in a cross-sectional study in the University Hospitals Munich, Freiburg, Berlin, Düsseldorf, Zurich, Basel, Berne, and the Cantonal Hospital St. Gallen (N=150). The goal of this project is that symptom assessment becomes a standard component of clinical practice (to promote the early detection and treatment of symptoms) and research.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* able to read and write German
* diagnosed with vulvar neoplasms
* treated with vulval surgery during the prior six month

Exclusion Criteria:

* cognitive impaired
* concurrently under psychiatric treatment or terminally ill

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with vulvar intraephitelial neoplasia or vulvar cancer following vulvar surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (4):
  - University Hospital Berlin, Berlin
  - University Hospital Dusseldorf, Düsseldorf
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Munich, Munich
- Switzerland (4):
  - University Hospital Basel, Basel
  - University Hospital Berne, Bern
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

REFERENCES:
- [Result] Senn B, Mueller MD, Cignacco EL, Eicher M. Period prevalence and risk factors for postoperative short-term wound complications in vulvar cancer: a cross-sectional study. Int J Gynecol Cancer. 2010 May;20(4):646-54. doi: 10.1111/IGC.0b013e3181d92723. PMID 20686386
- [Derived] Senn B, Eicher M, Mueller MD, Hornung R, Fink D, Baessler K, Hampl M, Denhaerynck K, Spirig R, Engberg S. A patient-reported outcome measure to identify occurrence and distress of post-surgery symptoms of WOMen with vulvAr Neoplasia (WOMAN-PRO) - a cross sectional study. Gynecol Oncol. 2013 Apr;129(1):234-40. doi: 10.1016/j.ygyno.2012.12.038. Epub 2013 Jan 3. PMID 23290987